CLINICAL TRIAL: NCT06740344
Title: Neonatal Mask Seal; a Randomised Controlled Trial of Two-handed Versus One-handed Hold for Delivering Positive-pressure Ventilation With a Facemask in Preterm and Term Infants: The NeoSeal Study
Brief Title: Neonatal Mask Seal; a Two-handed Versus One-handed Approach: The NeoSeal Study
Acronym: NeoSeal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EC36.2024
Record Dates: First submitted 2024-11-21; First posted 2024-12-18 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Neonatal Intensive Care
Keywords: Neonatology; Facemask ventilation; Face mask ventilation; Mask hold; One-handed mask hold; One-handed hold; Mask leak

STUDY DESIGN:
Intervention Model Description: Parallel group randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: This is an unblinded study as it is not possible to blind the provider to the type of mask hold. However, the operators will be blinded to the respiratory function monitor measurements feedback. This will be achieved by obscuring the colour sensor with brown, opaque tape and covering the Monivent screen. The outcome assessor will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: Two-handed facemask hold (Experimental): Two-handed mask hold technique while giving facemask ventilation, with another operator designated to deliver positive inspiratory pressure (PIP) via the T-piece. The operators may be any member of the neonatal team, who have undergone Neonatal Resusctiation Programme (NRP) certification. Standardised mask size and shape for gestation and weight, as per local policy, will be used.
  Interventions: Procedure: Two-handed facemask hold
- Control: One-handed facemask hold (Placebo Comparator): One-handed mask hold technique while giving facemask ventilation, with the same operator holding the mask and delivering positive pressure ventilation (PPV) via the T-piece.
  Interventions: Procedure: Control: One-handed facemask hold

INTERVENTIONS:
Procedure: Two-handed facemask hold — Two-handed mask hold technique while giving facemask ventilation, with another operator designated to deliver PIP via the T-piece.
  Arms: Intervention: Two-handed facemask hold
Procedure: Control: One-handed facemask hold — One-handed mask hold technique while giving facemask ventilation, with the same operator holding the mask and delivering PPV via the T-piece.
  Arms: Control: One-handed facemask hold

SUMMARY:
When babies can't breathe effectively, we can use a facemask to give them breaths and oxygen. The mask can be held with one or two hands, depending on the preference of the doctor. Both types of mask holds are recommended in international guidelines, but it is unclear which one is better for the baby. If a lot of air is leaking around the mask, it means that the baby is not getting the full breathing support that the healthcare providers are trying to give. There currently is not enough evidence to say which type of hold is better to reduce this potential leaking of air.

In this study, the investigators will compare two different ways of holding a mask on a baby's face to help them breathe. Each baby will be randomly allocated to either a one-handed or a two-handed mask hold, and the investigators will measure how much air leaks out around the mask during each breath. Any baby in the neonatal unit may be included in this study.

DETAILED DESCRIPTION:
This study will compare the measured leak in mask ventilation delivered by a healthcare professional in the neonatal team, using a one-handed versus a two-handed hold with a standardised mask size and shape. This is to assess the two-handed technique as a potential first-line approach in neonatal bag-mask ventilation.

The handholds will be assessed by a randomised controlled trial, with the two-handed hold as the intervention and the one-handed hold as the control.

The population that will be studied is neonates in the neonatal intensive care unit (NICU), at any gestation, who the clinical team have decided to intubate.

A member of the research team, who will provide an out-of-hours on call service, will attend the event. The relevant outcomes will be measured by the Monivent Neo100, which will be set up by the research team. Standardised masks, as used per local protocol, will be used, with the sensor module placed between that and the T-piece with an adaptor.

The outcomes will assess the effectiveness of both the intervention and control, including ventilation parameters recorded by the Monivent Neo100 and the clinical stability of the patient. The primary outcome of this study is the percentage mask leak.

A research team member will record data for primary and secondary outcome. The event will be filmed for post-hoc video analysis.

The outcome assessor will be blinded to the group allocation.

This research project will take place over 24 months, with an interim analysis to ensure recruitment is projected to achieve sample size.

ELIGIBILITY:
Inclusion Criteria:

* All term and preterm neonates in the neonatal unit who the clinical team have decided to intubate, with or without pre-medication and who require mask ventilation prior to intubation attempt.

Exclusion Criteria:

* Neonates with a congenital malformation that would impact mask seal will not be included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mask leak | Over a maximum of 20 minutes
  Mask leak percentage, as measured by the Monivent Respiratory Function Monitor (RFM).
  Collected over a minimum of 5 breaths. Maximum of 2 episodes of facemask ventilation will be collected, with values averaged.

SECONDARY OUTCOMES:
Lowest oxygen saturation | Over a maximum of 20 minutes
  Lowest oxygen saturation detected on the bedside clinical monitoring (Philips Intellivue MX800) during the period of facemask ventilation, recorded by a member of the research team.
Highest supplemental FiO2 used during facemask ventilation | Over a maximum of 20 minutes
  Highest percentage FiO2 used during the period of facemask ventilation, as indicated by the set dial on the Neopuff.
Positive inspiratory pressure during facemask ventilation | Over a maximum of 20 minutes
  Positive inspiratory pressure used during the period of facemask ventilation, as measured by the Monivent Neo100 respiratory function monitor.
Percentage of obstructed breaths during facemask ventilation | Over a maximum of 20 minutes
  Percentage of obstructed breaths during the period of facemask ventilation, as measured by the Monivent Neo100 respiratory function monitor.
Tidal volume during facemask ventilation | Over a maximum of 20 minutes
  Measured tidal volume during the period of facemask ventilation, as measured by the Monivent Neo100 respiratory function monitor.
Number of times facemask position is adjusted during facemask ventilation | Over a maximum of 20 minutes
  Number of times clinical team needs to adjust mask position during the period of facemask ventilation.
Duration of facemask ventilation | Over a maximum of 20 minutes
  Time duration of facemask ventilation
Crossover to other handhold | Over a maximum of 20 minutes
  If allocated two-handed hold: Number of times clinical team elect to switch to one-handed hold.
  If allocated one-handed hold: Number of times clinical team elect to switch to two-handed hold.
User opinion of mask hold | Over a maximum of 20 minutes
  Survey of operator opinions about mask hold used, and their usual preference.
Lowest heart rate | Over a maximum of 20 minutes
  Lowest heart rate detected on the bedside clinical monitoring (Philips Intellivue MX800) during the period of facemask ventilation, recorded by a member of the research team.

CONTACTS AND LOCATIONS:
Locations (1):
- The National Maternity Hospital Dublin, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: No
Data will be pseudononymised and will be presented/shared only as collated values, as opposed to individual results.

REFERENCES:
- [Background] Newborn Life Support. J. Fawke et al. Resuscitation Council UK. May 2021.
- [Background] Shah D, Tracy MB, Hinder MK, Badawi N. One-person versus two-person mask ventilation in preterm infants at birth: a pilot randomised controlled trial. BMJ Paediatr Open. 2023 Feb;7(1):e001768. doi: 10.1136/bmjpo-2022-001768. PMID 36746525
- [Background] Tracy MB, Klimek J, Coughtrey H, Shingde V, Ponnampalam G, Hinder M, Maheshwari R, Tracy SK. Mask leak in one-person mask ventilation compared to two-person in newborn infant manikin study. Arch Dis Child Fetal Neonatal Ed. 2011 May;96(3):F195-200. doi: 10.1136/adc.2009.169847. Epub 2010 Nov 11. PMID 21071683
- [Background] Murray A, Beechinor T, Livingstone V, Dempsey E. Two hands are better than one: Positive pressure ventilation in a preterm neonatal manikin model. Acta Paediatr. 2024 May;113(5):989-991. doi: 10.1111/apa.17156. Epub 2024 Feb 22. No abstract available. PMID 38389164
- [Background] Wood FE, Morley CJ. Face mask ventilation--the dos and don'ts. Semin Fetal Neonatal Med. 2013 Dec;18(6):344-51. doi: 10.1016/j.siny.2013.08.009. Epub 2013 Sep 14. PMID 24041823
- [Background] Weiner GM, Zaichkin J. Updates for the Neonatal Resuscitation Program and Resuscitation Guidelines. Neoreviews. 2022 Apr 1;23(4):e238-e249. doi: 10.1542/neo.23-4-e238. PMID 35362042
- [Background] O'Currain E, O'Shea JE, McGrory L, Owen LS, Kamlin O, Dawson JA, Davis PG, Thio M. Smaller facemasks for positive pressure ventilation in preterm infants: A randomised trial. Resuscitation. 2019 Jan;134:91-98. doi: 10.1016/j.resuscitation.2018.12.005. Epub 2018 Dec 17. PMID 30572069